CLINICAL TRIAL: NCT06180291
Title: Impact of a Screening and Early Intervention Program on the Functional Impact of Cerebral Palsy at 2 Years in Children at High Risk of Cerebral Palsy: a Prospective Comparative Multicenter Study.
Brief Title: EARLY Intervention in Parent-professional Cooperation in Cerebral Palsy
Acronym: PRECOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 69HCL22_0862
Record Dates: First submitted 2023-10-23; First posted 2023-12-22 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy
Keywords: early intervention program; functional impact; cerebral palsy; children
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Prospective multicenter comparative non-randomized study evaluating the effectiveness of a new management strategy for children at high risk of cerebral palsy compared to the management of the control group.
  The research will take place in 8 centers, 4 centers offering early intervention (Lyon Croix-Rousse, Lyon Hôpital Femme-Mère-Enfant, Montpellier, Nîmes), and 4 centers not offering standardized early intervention (Toulouse neonatal care unit, Toulouse pediatric intensive care unit, Chambéry and Annecy). The control centers were recruited on the basis of common characteristics of neonatology level of care and active queue.
  Each center will consecutively include newborns during the neonatology stay. The study will compare the intervention group composed of children cared for in intervention centers to the control group composed of children cared for in control centers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): PRECOP group: screening and early treatment. CAMSP (Centre d'Action Médico-Sociale Précoce) orientation upon discharge from neonatology for immediate follow-up according to PRECOP protocol: early multidisciplinary care, with targeted objectives according to the child's needs.
  Interventions: Other: PRECOP program
- Control group (No Intervention): Standard of care group: in the control centers, care includes specialized consultations organized by the perinatal network with a hospital and/or community pediatrician belonging to the network until the child is 2 years old. Cerebral palsy screening is based on clinical examination.

INTERVENTIONS:
Other: PRECOP program — PRECOP program is the first program combining early detection of cerebral palsy with implementation of early interventions following the latest international recommendations (multidisciplinary program at home, with the possibility of intensive courses, coaching parental, in the first 2 years of life).
  This comprehensive monitoring is implemented as soon as the infant arrives at home, by a multidisciplinary team and continues during the child's first 2 years. It includes:
  * Follow-up organized primarily at home
  * Monitoring of psychomotor development
  * Screening for possible cerebral palsy
  * Comprehensive support for the child's development: weight, diet, sleep...
  * Reeducation, implementation of SMART type objectives (Specific, Measurable, Achievable, Achievable, Timely defined) determined with parents
  * Creation of equipment if necessary: early seating installation in particular
  * Parental support and guidance for optimizing early care
  * Parental psychological support.
  Arms: Intervention group

SUMMARY:
Cerebral Palsy (CP) is the most common motor disability in children. It is due to damage that occurs during brain development in the fetus or infant. Early treatment (before 2 years) will allow the child to promote brain plasticity to compensate for the effects of the lesion and reduce the severity of CP. The goals of early intervention are to increase motor, cognitive and communication skills, prevent complications and provide parental support. Most authors agree to recognize the benefit of early care by emphasizing home intervention programs with active parental participation. To date, no recommendations exist in France for the management of cerebral palsy in children under the age of two. It is therefore necessary to conduct scientific studies in this population.

Based on published international studies, the PRECOP program (PREcoce intervention in parent-professional COoperation in Cerebral Palsy) consists of individualized care adapted to the specific needs of each child, from the arrival of the infant at home, by a multidisciplinary team during the child's first two years.

ELIGIBILITY:
Inclusion Criteria:

* New born presenting on transfontanellar ultrasound and confirmed on brain MRI (magnetic resonance imaging) at least one of the following brain lesions at high risk of cerebral palsy :

  * Stage 3 intraventricular hemorrhage, requiring at least 2 subtractive lumbar punctures and/or the establishment of a ventriculoperitoneal bypass
  * Stage 4 intraventricular hemorrhage
  * Periventricular leukomalacia : extensive unilateral or bilateral
  * Sequelae of perinatal anoxo-ischemic encephalopathy
  * Extensive neonatal stroke
* Less than 3 months old (corrected age in case of prematurity)
* Hospitalized in neonatology or hospitalized in pediatric intensive care unit or within two months following return home (follow-up visit after initial hospitalization)
* Affiliate to social security
* Parental or legal representative consent to participate in the study (free and informed written consent)

Exclusion Criteria:

* Children who have had an Antenatal Diagnosis of a pathology causing fear of the onset of developmental delay
* Children presenting with a congenital pathology with neonatal revelation, whether of metabolic, genetic or malformative origin
* Palliative care offered by the neonatology team (LATA: Limitation and Discontinuation of Active Therapeutics)
* Children participating simultaneously in another screening and early care program (excluding the COCON program (Soins préCOces et COordonnés du Nouveau-né vulnérable))

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Score of the Total Motor Index at PDMS-3 scale (Peabody Developmental Motor Scales). | 24 months
  Score of the Total Motor Index at PDMS-3 scale (Peabody Developmental Motor Scales).The Total Motor Index results from the combination of Gross Motor Index and Fine Motor Index scores at PDMS-3. The functional impact of cerebral palsy at 2 years is assessed by the PDMS-3 at 24 months of age will be estimated in each of the two groups by a mean value with a 95% confidence interval.

SECONDARY OUTCOMES:
Motor development | 24 months
  The assessment of motor development will be completed by taking the Global Functional Motor Assessment (EMFG) Scale ranging from 0 to 3, with 3 being the best.
Cognitive development | 24 months
  Cognitive development will be measured by the Ages and Stages Questionnaire (ASQ)
Nutritional development | 24 months
  Nutritional development will be assessed by the Montreal Children's Hospital (MCH) Eating Scale Scale ranging from 1 to 7, with the best score depending on each item.
Development of Production Language in French (DLPF) questionnaire | 24 months
  The development of communication and language will be assessed through the Development of Production Language in French (DLPF) questionnaire
Early relational problems | 24 months
  Early relational problems will be detected by Modified Checklist for Autism in Toddlers (M CHAT)
Parental stress | 24 months
  Parental stress will be measured at 24 months of the child by the Parental Stress Scale (ESP for "Echelle de Stress Parental" in french).
  Scale ranging from 1 to 5, with the best score depending on each item.
Implemented intervention and fidelity to the planned intervention at the center level | through study completion, an average of 42 months
  Number of professionals trained and profile of professionals, human, material and organizational resources mobilized.
Intervention implemented and fidelity to the planned intervention at the patient level | through study completion, an average of 42 months
  Number of components of the intervention received, compliance with the frequency of interventions and deadlines in relation to the course planned to achieve the child's objectives.
Parental adherence | through study completion, an average of 42 months
  Parental adherence to the recommendations given in the PRECOP program evaluated according to the number of sessions not carried out or canceled by the parents.
Acceptability of the intervention | through study completion, an average of 42 months
  Acceptability from the parents' and professionals point of view, assessed by a questionnaire constructed for the study.
Program transferability using PIET model: Population, Intervention, Environment, Transfer | through study completion, an average of 42 months
  Assessing whether PRECOP programm can be transferred from the "primary context" (the context of the intervention as it was performed in the original study) to the "target context" (the context that the intervention is aimed at being performed in) using PIET model : Population, Intervention, Environment, Transfer.
Cost ratio impact | 12, 24 and 36 months
  Differential cost ratio resulting from the PRECOP strategy compared to the management of the control group.
Annual cost impact | 12, 24 and 36 months
  Average annual cost of support for the financier depending on the pricing methods.
Budgetary impact | 12, 24 and 36 months
  Estimating annual net budget up to 3 years according to trial data, literature and expert opinion.

CONTACTS AND LOCATIONS:
Overall Officials: Virginie MOURON, MD, Principal Investigator — Service de Réanimation Néonatale, Hôpital de la Croix-Rousse, Hospices Civils de Lyon
Locations (8):
- France (8):
  - CH de Annecy, Annecy
  - Service de Réanimation et médecine néonatale, Chambéry
  - Service de Réanimation Néonatale, Hôpital de la Croix-Rousse, Hospices Civils de Lyon, Lyon
  - Service de néonatologie et de réanimation néonatale, Hôpital Femme Mère Enfant, Hospices Civils de Lyon, Lyon
  - Service de néonatologie et de réanimation néonatale, CHU Saint-ELOI, Montpellier
  - Service de néonatologie et de réanimation néonatale, Hôpital Universitaire Carémeau, Nîmes
  - Service de réanimation pédiatrique, Hôpital des enfants, Toulouse
  - Service de néonatologie, Hôpital des enfants, Toulouse

IPD SHARING:
Plan to Share IPD: No